CLINICAL TRIAL: NCT00259389
Title: Directly Observed Therapy (DOT) in HIV-1 Infected Adolescents
Brief Title: Directly Observed Therapy for HIV Infected Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Pediatric AIDS Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PACTG P1036B; 10044 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 2005-11-28; First posted 2005-11-29 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: HIV Infections
Keywords: Treatment Experienced; Adherence; Compliance; Directly Observed Therapy; DOT; Treatment Naive
MeSH Terms: conditions — HIV Infections; Patient Compliance; Directly Observed Therapy

INTERVENTIONS:
Behavioral: Directly observed therapy (DOT)

SUMMARY:
Adherence to a doctor-prescribed anti-HIV drug regimen is crucial in the management of HIV infection. In previous studies with tuberculosis patients, directly observed therapy (DOT), a strategy in which patients are observed while taking their medications, has been proven useful in increasing patient adherence. The purpose of this study is to determine the effectiveness of a new DOT strategy in HIV infected adolescents who have had difficulty adhering to anti-HIV drug regimens or regimens to prevent opportunistic infections (OIs) in the past.

DETAILED DESCRIPTION:
For HIV infected people, control of HIV infection is best achieved by adhering to the highly active antiretroviral therapy (HAART) regimen prescribed by their doctors. Poor adherence to a HAART regimen leads to clinical failure and the development of resistance. Many HIV infected adolescents have difficulty adhering to their prescribed anti-HIV regimens or OI prophylaxis; often, they cite forgetting to take their medications as the reason for poor adherence. This is a pilot study of using DOT and assessing adherence during DOT in HIV infected adolescents who have had difficulty adhering to HAART regimens in the past. The purpose of this study is to evaluate the efficacy in increasing patient adherence and the feasibility of using DOT among HIV infected adolescents.

This study will last 24 weeks. For the first 2 weeks of the study, DOT will be provided 7 days a week at the study site; participants will visit the study site daily and will be observed taking their medication. For the next 6 weeks, the frequency of DOT will be reduced from 7 days a week to 5 days a week. Based on adherence from Weeks 4 to 8, each participant will be recommended to continue with a DOT strategy as follows:

* Adherence Level 1 (greater than 93%) - DOT 3 days a week
* Adherence Level 2 (86% to 93%) - DOT 5 days a week
* Adherence Level 3 (less than 86%) - DOT 7 days a week

Participants will decide whether to accept their DOT assignment and to continue in the study. At Week 12 and every 4 weeks thereafter, adherence will be assessed and DOT may be adjusted as follows:

* Adherence Level 1 - Reduce frequency of DOT. Those already receiving DOT 3 days a week stop DOT and start self-administered therapy.
* Adherence Level 2 - Keep same frequency of DOT as the past 4 weeks.
* Adherence Level 3 - Increase frequency of DOT by one level, as described in previous list.

HAART will not be provided by this study, so participants must have access to their HAART medications coordinated separately through the study site. Participants who are taking medication requiring twice-daily dosing will self-administer their second doses.

There will be 7 study visits; they will occur at study entry and every 4 weeks thereafter. Medical history will occur at study entry. At every visit, participants' adherence to their regimens will be assessed, and they will also be interviewed by a social worker about their use of support services. Participants will undergo several assessments at study entry and Weeks 12 and 24 to determine participant confidence, beliefs about medicine, severity of depression, feelings of hopelessness, coping responses, and emotional and behavioral problems. Blood collection will occur at study entry and Weeks 8, 12, and 24. When participants successfully complete their prescribed courses of DOT or elect to discontinue DOT, they will again be interviewed by study staff.

ELIGIBILITY:
Inclusion Criteria:

* Infected with HIV after age 12
* Initiating, continuing, changing, or reinitiating a daily or twice-daily HAART regimen AND have demonstrated adherence problems (less than 85% of prescribed doses taken, as clinically disclosed, on 2 consecutive occasions at least 1 month apart). More information on this criterion can be found in the protocol.
* Able and willing to swallow medication
* Have access to HAART
* Parent or guardian willing to provide informed consent, if applicable
* Willing to use acceptable forms of contraception

Exclusion Criteria:

* Clinically significant diseases other than HIV infection or clinically significant findings during screening or physical examination that, in the opinion of the investigator, would require much closer follow-up and frequent monitoring than would be generally done for other HIV infected patients of comparable age
* HAART regimens that include medications taken more often than twice-daily
* Investigational agents (HAART or other medications) administered as part of other clinical trials
* Pregnant or breastfeeding

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2006-04; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Proportion of completed directly observed therapy (DOT) facilitator-participant interactions, among all scheduled interactions, for each participant during the second 4-week period on study
number and proportion of participants who were able to complete the recommended duration of DOT

SECONDARY OUTCOMES:
Subject satisfaction with DOT, assessed by the Exit Survey Instrument
cost of implementing DOT per participant
effective ratio of DOT facilitators to participants, determined by the calculation of actual time spent by each DOT facilitator
reproducibility of DOT implementation across sites and participants' adherence to DOT interactions and ability to complete the prescribed duration of DOT, compared across sites
adherence for each participant in the 4-week period prior to a study visit, determined at Weeks 8 and 12 by participant self-report and adherence to DOT interactions and by pill count and participant 4-week recall at Week 24
virologic outcomes, determined by the suppression of HIV-1 viral load at Weeks 8, 12, and 24
immunologic outcome, defined by a change in absolute CD4 count from baseline to Week 24
self-efficacy (confidence), assessed by Patient Assessment Tool - Part I and Beliefs About Medicine Scale
beliefs about highly active antiretroviral therapy (HAART), assessed by Beliefs About Medicine Scale
severity of depression experienced by each participant, assessed by Beck Depression Inventory (BDI)-II
hopelessness, assessed by Beck Hopelessness Scale (BHS)
emotional and behavioral problems, assessed by Youth Self Report (YSR)/Adult Self Report (ASR)
coping of each participant, assessed by Coping Responses Inventory (CRI)-Youth and CRI-Adult
perceived barriers to adherence, assessed at baseline and Weeks 12 and 24 by Patient Assessment Tool - Part I and Beliefs About Medication Scale
substance abuse, assessed at baseline and Weeks 12 and 24 by Patient Assessment Tool - Part II
sustainability of DOT benefits, assessed as the proportion of participants adherent at Week 24 among those who successfully complete the first 8 weeks of DOT and are taken off DOT at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Aditya Gaur, MD, Study Chair — Department of Infectious Disease, St. Jude Children's Research Hospital
Locations (6):
- United States (6):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Los Angeles County Medical Center/USC, Los Angeles, California
  - UCSD Mother, Child & Adolescent HIV Program, San Diego, California
  - Childrens Hospital of Michigan, Detroit, Michigan
  - University of Rochester Medical Center, Rochester, New York
  - St. Jude Childrens Research Hospital, Memphis, Memphis, Tennessee

REFERENCES:
- [Background] Martinez J, Bell D, Camacho R, Henry-Reid LM, Bell M, Watson C, Rodriguez F. Adherence to antiviral drug regimens in HIV-infected adolescent patients engaged in care in a comprehensive adolescent and young adult clinic. J Natl Med Assoc. 2000 Feb;92(2):55-61. PMID 10800292
- [Background] Mitty JA, Stone VE, Sands M, Macalino G, Flanigan T. Directly observed therapy for the treatment of people with human immunodeficiency virus infection: a work in progress. Clin Infect Dis. 2002 Apr 1;34(7):984-90. doi: 10.1086/339447. Epub 2002 Feb 27. PMID 11880965
- [Background] Murphy DA, Sarr M, Durako SJ, Moscicki AB, Wilson CM, Muenz LR; Adolescent Medicine HIV/AIDS Research Network. Barriers to HAART adherence among human immunodeficiency virus-infected adolescents. Arch Pediatr Adolesc Med. 2003 Mar;157(3):249-55. doi: 10.1001/archpedi.157.3.249. PMID 12622674
- [Background] Wohl AR, Garland WH, Squires K, Witt M, Larsen R, Kovacs A, Hader S, Weidle PJ. The feasibility of a community-based directly administered antiretroviral therapy program. Clin Infect Dis. 2004 Jun 1;38 Suppl 5:S388-92. doi: 10.1086/421401. PMID 15156427
- [Result] Garvie PA, Flynn PM, Belzer M, Britto P, Hu C, Graham B, Neely M, McSherry GD, Spector SA, Gaur AH; Pediatric AIDS Clinical Trials Group (PACTG) P1036B Team. Psychological factors, beliefs about medication, and adherence of youth with human immunodeficiency virus in a multisite directly observed therapy pilot study. J Adolesc Health. 2011 Jun;48(6):637-40. doi: 10.1016/j.jadohealth.2010.09.014. Epub 2010 Dec 18. PMID 21575827